CLINICAL TRIAL: NCT01902849
Title: The Influence of Anesthetic Technique on Interleukin Plasma Level in Colorectal Cancer Surgery - TIVA vs Inhalation Anesthesia
Brief Title: Anesthetic Technique on Immune Response in Colorectal Cancer
Acronym: T-IL-Co-ReCa
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Margarit Simona, senior lecturer, consultant in anesthesia and intensive care, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: TICC
Record Dates: First submitted 2013-07-13; First posted 2013-07-18 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Colorectal Neoplasms
Keywords: intravenous anesthesia; inhalational anesthesia; interleukins; colorectal surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — The collected blood samples are centrifuged at 2500 rpm / min for 10 minutes and the resulting plasma is stored at -70 °
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1 - TIVA-TCI: * include 35 patients with colorectal cancer undergoing surgery
  * anaesthesia is induced and maintained with total intravenous target-controlled infusion ( TIVA-TCI) of propofol and remifentanil.
  * for propofol initial target plasma concentration (Cp) is set to 4 micrograms/ml (modified Marsh model)( Base Primea™, Fresenius, France) and then adjusted in steps 0.2 micrograms/ml to maintain the BIS values between 40-55 during surgery.
  * for Remifentanil initial Cp is set at induction at 4 ng/ml and then the Cp is maintained between 3-8 ng/mL(increments of 0.5 ng/ml in case of inadequate anesthesia).
  * intervention:blood sampling for IL measurement
  Interventions: Other: blood sampling for IL measurement
- Group II- ISOFLURANE: * include 35 patients with colorectal cancer undergoing surgery
  * anesthesia is induced with propofol bolus 1,5-2 mg/kg and remifentanil TCI mode (Minto model) (Base Primea™, Fresenius, France) with an initial Cp 4 ng/ml
  * maintenance of anesthesia is achieved with isoflurane 1-1.5 MAC in order to maintain the BIS value between the values of 40-55 and remifentanil TCI with Cp between 3-8 ng/mL (increments of 0.5 ng/ml in case of inadequate anesthesia)
  * intervention:blood sampling for IL measurement
  Interventions: Other: blood sampling for IL measurement

INTERVENTIONS:
Other: blood sampling for IL measurement — Blood sampling to determine interleukins IL6 , IL10 plasma levels are drawn at the following moments:
  * T0- before the induction of anesthesia (venous cannula insertion time)
  * T1- after induction but before starting surgery
    * In the group I (TIVA -TCI) when the plasma concentration of propofol is 3-3.5 ng/ml
    * In group II (ISOFLURANE) when concentration of isoflurane in exhaled air (Et Isoflurane) is between 0.3-0.5%
  * T2, T3- at 2 and 24 hours after surgery

SUMMARY:
Knowing the fact that the anesthetic substances can alter the immune response during the surgery, the purpose of the study is to evaluate the influence of two general anesthetic techniques - inhalation vs. total intravenous anesthesia on the immune response in patient with colorectal surgery for neoplastic disease, evaluated by the plasma level of the interleukins 6 and 10(IL6, IL10).

DETAILED DESCRIPTION:
Introduction

Several factors are contributing to perioperative immunosuppression such as: surgery itself, general anesthesia. In vivo and in vitro studies have shown that anesthesia itself may alter the immune response either by direct effect on immune cells (such as natural killer and T helper) ) or indirectly by the influence of anesthetic substances on pro (IL-1, IL-6, tumor necrosis factor alpha ) and anti-inflammatory ( IL-4, IL-10) cytokines release.

The study aims to evaluate the influence of two general anesthetic techniques inhalation versus total intravenous anesthesia- target controlled infusion (TIVA-TCI) on the immune response in patient with colorectal surgery for neoplastic disease, evaluated by the plasma level of the interleukins IL6, IL10.

Study group:

- patients admitted to the Surgical Clinic of the Regional Institute of Gastroenterology and Hepatology Prof Dr Octavian Fodor, undergoing open surgery for colorectal cancer (right/left colectomy, colorectal resection).

After obtaining written informed consent 70 ASA physical status I-III patients scheduled for colorectal cancer resection are randomly allocated to 2 groups of study by computer randomization:

* group I, TIVA-TCI (n=35 patient) receive total intravenous-target controlled infusion anesthesia with propofol and remifentanil
* group II (ISOFLURANE) (n=35 patients) receive inhalatory anesthesia with isoflurane and remifentanil

Methods:

* Premedication with midazolam 7.5 mg orally 30 min before surgery in all patients.
* On arrival in the operating room a venous cannula is inserted and a blood sample for interleukin measurement is performed. This cannula is designated for fluid administration during anesthesia and for blood sampling for subsequent interleukin measurements. A second cannula is inserted for the administration of anesthetic substances.

In group I (TIVA-TCI):

* anesthesia is induced with a target-controlled infusion (TCI) of propofol with an initial target plasma concentration (Cp) of 4 micrograms/ml (modified Marsh model)( Base Primea™, Fresenius, France), adjusted in steps 0.2 micrograms/ml to maintain the BIS values between 40-55 during surgery.
* propofol infusion stops at the end of surgery before the last 2 stitches.

In group II (ISOFLURANE):

* anesthesia is induced with propofol bolus 1,5-2 mg/kg.
* maintenance of anesthesia is achieved with isoflurane 1-1.5 MAC in order to maintain the BIS value between the values of 40-55.
* isoflurane administration cease before the last 2 stitches.

In both groups:

* remifentanil TCI mode (Minto model) (Base Primea™, Fresenius, France) is used for analgesia, with an initial Cp of remifentanil set at 4 ng/ml at induction, and a Cp between 3-8 ng/mL during maintenance(increments of 0.5 ng/ml) depending on the painful moments of surgery and the patient's analgesic needs assessed by changes in heart rate, blood pressure (more than 20% of the previous value of induction), sweating, tearing.
* remifentanil infusion ceases after suturing the wound.
* muscle relaxation is achieved with atracurium, 0.5-0.6 mg/kg at induction, and further maintained on top up doses as needed. At the end of surgery the residual neuromuscular blockade is reversed with atropine 0.02mg/kg and neostigmine 0.0 5mg/kg.
* the lungs are ventilated with an air/oxygen mixture.

Postoperative analgesia:

* morphine patient controlled analgesia(PCA ) with boluses of 1 mg to 5 min interval to maintain the VAS ˂ 4 on 10-point visual analogue scale (VAS). The first dose of morphine 0.1 mg/kg is administered 40 minutes before completing the surgery.
* in addition to morphine, is given paracetamol intravenous, 1g every 8 hours. The first dose of paracetamol is administered intra-operatively before the end of surgery.

Monitoring:

1. Intraoperative:

   * ASA basic monitoring: continuous monitoring ECG, heart rate (HR), arterial blood pressure (BP), pulse oximetry (SpO2), CO2 concentration in expired gases (Et CO2), concentration of isoflurane in exhaled gases (Et Iso), minimum alveolar concentration (MAC) of isoflurane, and core temperature.
   * depth of anesthesia - bispectral index (BIS) (BIS Vista -Aspect Medical System, USA).

   Systolic, diastolic blood pressure and HR are recorded every minute at induction time and every 5 minutes after endotracheal intubation, until the end of surgery.

   Hypotension (defined as a decrease of mean arterial blood pressure by over 20% of baseline values) is treated with higher rate of infusion solutions and intravenous boluses of ephedrine 5 mg.

   Inadequate anesthesia (hypertension, tachycardia, lacrimation, sweating) is treated by adjusting the remifentanil infusion as previously mentioned.
2. Postoperative:

   * opioid analgesic requirement in the first 24 hours
   * pain score on the visual analog scale (VAS 0-10)in the first 24 hour
   * incidence of postoperative nausea and vomiting episodes requiring the administration of antiemetic drug (metoclopramide 20 mg or ondansetron 4 mg)

Blood sampling to determine interleukins IL6 , IL10 plasma levels are drawn at the following moments:

* T0- before the induction of anesthesia (venous cannula insertion time)
* T1- after induction but before starting surgery:

  * in group I (TIVA -TCI) when the plasma concentration of propofol is 3-3.5 micrograms/ml
  * in group II (ISOFLURANE) when concentration of isoflurane in exhaled air (Et Isoflurane) is between 0.3-0.5%
* T2, T3 - at 2 and 24 hours after surgery

The collected blood samples are centrifuged at 2500 rpm / min for 10 minutes and the resulting plasma is stored at -70 ° C until the interleukins assay is performed.

If intraoperatively is revealed local extension of colorectal cancer (tumor invades adjacent organs) or distant metastasis the patient is excluded from the study.

Data collection is done longitudinally prospective, for each patient the following variable are registered:

* quantitative: - weight, plasmatic or brain concentration of the anesthetics used in TIVA-TCI mode, BIS value, plasmatic concentration of the interleukins on 4 intra- and post-operatory moments, the duration of the surgery and anesthesia, number of episodes of nausea and vomiting, opioid analgesic requirement.
* qualitative: ASA score, sex, post-operatory pain score (VAS) Collected data are introduced in a database using the Excel Office programme.

The statistical analysis will be performed using the SPSS 16.0 software (SPSS Inc Chicago, IL, USA). Quantitative variables will be expressed as mean ± SD, and qualitative variables as absolute and relative frequencies. Given multiple measurements at different time intervals, area under curve (AUC) is calculated for each IL and the results will be compared between groups.A p less 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years with ASA physical status I-III.
* colorectal cancer patients with no sign of local invasion (adjacent organs) and distant metastasis revealed by imaging studies
* surgery performed by the same surgical team

Exclusion Criteria:

* ASA physical status IV patients
* hepatic and renal impairment
* diabetes or other endocrine disorders
* obesity (BMI 30 kg/m2)
* immune disorders or immunosuppressive therapy
* steroid treatment in the last 6 months
* asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with colorectal neoplasms
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
measurement of interleukins IL6 and IL 10 plasmatic level | -before anesthesia induction (T0 time)
  -once the intravenous cannula is inserted
measurement of interleukins IL6, IL10 plasmatic level | after anesthesia induction but before surgical incision (T1)
  * in group I (TIVA-TCI) when plasma concentration of propofol is 3-3.5 micrograms/ml
  * in group II (ISOFLURANE) when concentration of isoflurane in exhaled gases (Et iso) is between 0.3-0.5 %
measurement of interleukins IL6 and IL10 plasmatic level | 2 hours postoperatively (T2)
measurement of interleukins IL6 and IL 10 plasmatic level | 24 hours postoperatively (T3)

SECONDARY OUTCOMES:
total opioid analgesic dose (mg) | for the first 24 hours postoperatively

OTHER OUTCOMES:
Pain score on the visual analog scale (VAS 0-10) | for the first 24 hour postoperatively
  at 15, 30 minutes post surgery 6, 12, 18, 24 hours postoperatively
incidence of postoperative nausea and vomiting episodes requiring antiemetic medication | for the 24 hours postoperatively
total opioid dose of remifentanil (mg ) used during surgery | an average 3 hours
  total dose (mg) of remifentanil administered in TCI mode during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Simona C Margarit, lecturer, Principal Investigator — University of Medicine and Pharmacy Iuliu Hatieganu
Locations (1):
- University of Medicine and Pharmacy Iuliu Hatieganu; Regional Institute of Gastroenterology and Hepatology Prof Dr Octavian Fodor, Cluj-Napoca, Romania

REFERENCES:
- [Background] Ke JJ, Zhan J, Feng XB, Wu Y, Rao Y, Wang YL. A comparison of the effect of total intravenous anaesthesia with propofol and remifentanil and inhalational anaesthesia with isoflurane on the release of pro- and anti-inflammatory cytokines in patients undergoing open cholecystectomy. Anaesth Intensive Care. 2008 Jan;36(1):74-8. doi: 10.1177/0310057X0803600113. PMID 18326136
- [Derived] Margarit SC, Vasian HN, Balla E, Vesa S, Ionescu DC. The influence of total intravenous anaesthesia and isoflurane anaesthesia on plasma interleukin-6 and interleukin-10 concentrations after colorectal surgery for cancer: a randomised controlled trial. Eur J Anaesthesiol. 2014 Dec;31(12):678-84. doi: 10.1097/EJA.0000000000000057. PMID 24614619